CLINICAL TRIAL: NCT06572059
Title: The Relationship Between Upper Extremity Motor Imagery Ability, Upper Extremity Functional Skills and Quality of Life in Patients With Multiple Sclerosis
Brief Title: Upper Extremity Motor Imagery Functional Skills and Quality of Life in Patients With Multiple Sclerosis
Acronym: MotorImagery
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Asistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: KahramanmarasSUI
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis; Upper Extremity Problem; Quality of Life; Image, Body; Motor Activity
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study/1(Assesments will be done for once): It will consist of individuals with MS (>18years old). who were followed up in the Multiple Sclerosis clinic of the Neurology Department of Kahramanmaraş Sutcu Imam University (KSU) Health Practice and Research Hospital. Patients who meet the inclusion criteria will be evaluated using the following parameters, respectively:
  * EDSS score (patient reports recorded by the physician will be used.)
  * Demographic information
  * Fatigue Severity Scale (FSS)
  * Beck Depression Inventory (BDI)
  * Kinesthetic and Visual Imagery Questionnaire (KVIQ)
  * Mental Chronometer Test (Nine-Hole Peg Test (DDPT) will be used.)
  * Jebson-Taylor Hand Function Test (JHEFT)
  * Manual Ability Test (MAM-36)
  * Multiple Sclerosis Impact Scale (MSIS-29) Assesments will be done for once.
  Interventions: Other: assesments for once
- healthy control/2 (Assesments will be done for once): It will consist of individuals with healthy volunteers with the similar age (>18years old).
  Healthy volunteers who meet the inclusion criteria will be evaluated using the following parameters, respectively:
  * EDSS score (patient reports recorded by the physician will be used.)
  * Demographic information
  * Fatigue Severity Scale (FSS)
  * Beck Depression Inventory (BDI)
  * Kinesthetic and Visual Imagery Questionnaire (KVIQ)
  * Mental Chronometer Test (Nine-Hole Peg Test (DDPT) will be used.
  * Jebson-Taylor Hand Function Test (JHEFT)
  * Manual Ability Test (MAM-36)
  * Multiple Sclerosis Impact Scale (MSIS-29) Assesments will be done for once.
  Interventions: Other: assesments for once

INTERVENTIONS:
Other: assesments for once — * EDSS score (patient reports recorded in the physician's record will be used.)
  * Demographic information
  * Fatigue Severity Scale (FSS)
  * Beck Depression Inventory (BDI)
  * Kinesthetic and Visual Imagery Questionnaire (KSVI)
  * Mental Chronometer Test (Nine-Hole Peg Test (DDPT)) will be used.)
  * Jebson-Taylor Hand Function Test (JHEFT)
  * Manual Ability Test (MAM-36)
  * Multiple Sclerosis Impact Scale (MSIS-29)

SUMMARY:
Multiple sclerosis (MS) is a chronic inflammatory and autoimmune disease of the central nervous system (CNS) characterised by axonal loss and demyelination. MS is characterized by myelin, oligodendrocyte and axon damage. MS progresses in a wide spectrum, with motor, sensory, autonomic and cognitive disorders depending on the area affected.

Upper extremity dysfunction is common in patients with MS (pwMS), too. 75% of pwMS have impaired ability to perform activities of daily living (ADL) and quality of life (QoL).

Motor imagery (MI) refers to the mental simulation of an action without physical intervention.

MS is also characterised by motor and cognitive symptoms. Cognitive impairment, seen in approximately 40-70% of patients, is mainly related to problems in attention, information processing speed, memory, cognitive and visual structure. MI refers to the mental simulation of an action without physical intervention, which can be classified as explicit or implicit. MI skill is linked to motor planning and execution skills. MI is related to the subconscious activation of motor systems that play a role not only in producing movement, but also in imagining actions, learning through observation, recognising tools, and also understanding other people's behaviour.The speed and quality of upper extremity functional skills in pwMS may be related to MI ability.

Health-related quality of life (HRQoL) is an individual's assessment of how a health problem and its treatment affect their ability to perform daily activities and roles. Research studies have shown that pwMS report lower QoL scores than healthy controls. Losses in upper extremity functional skills may affect the activities of daily living and work life in pwMS, leading to a decrease in their QoL. When evaluating MI ability in these patients, the patient's functional skills and cognitive status should also be taken into consideration.

It is thought that upper extremity MI skills may be negatively affected by impairments with the cognitive syptoms in pwMS. The aim of this study is to investigate the relationship between upper extremity MI ability, upper extremity functional skills and QoL in pwMS.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS), a chronic inflammatory disease of the central nervous system (CNS), is characterized by myelin, oligodendrocyte and axon damage.MS is a chronic disease with unpredictable clinical presentations, ranging from mild, infrequent relapses causing mild functional impairment to severe disability, including loss of independent walking or severe cognitive impairment.Upper limb dysfunction is common in patients with MS (pwMS). 75% of pwMS report difficulties performing bimanual tasks that affect their independence and ability to perform daily activities and quality of life (QoL). Such dysfunction is typically a combination of sensory, motor, and central deficits that occur proximally, distally, or throughout both upper limbs and may occur unilaterally or bilaterally.Upper extremity disability in pwMS can be found in the proximal or distal parts of the upper extremity. Distal upper extremity dysfunction is often referred to as impaired manual dexterity or hand dysfunction. Impaired sensory function, fatigue, loss of manual skills, and mobility are the most commonly reported symptoms in the first year of the disease in pwMS. It has also been reported that 75% of the population with MS at the level 6.5 according to the Expanded Disability Status Scale (EDSS) has impaired bimanual skills.

Motor imagery (MI) refers to the mental simulation of an action without physical intervention, which can be classified as explicit or implicit. Expilicit MI is defined as consciously imagining an action. This ability is assessed with Mental Chronometer (MK) and MI questionnaires. In implicit MI some tests such as mental rotation (MR) are applied to ensure that individuals can use their ability unconsciously. MI skills are related to motor planning and execution skills.MI supports motor learning and motor performance and is a useful strategy for neurorehabilitation. The mechanism of this imagery involves activating the same sensorimotor regions in the brain that are active during the physical completion of the movement, thus potentially strengthening and increasing synaptic connectivity for the regions involved in the movement. Areas involved in this activation include the primary motor cortex, basal ganglia, cerebellum, premotor cortex, supplementary motor area, parietal cortex, and prefrontal cortex. The corticospinal tract is activated during MI, an important indication that the imagery stimulates surrounding motor neurons and affects the cortex. These neural networks are activated during MI, strengthening connections and improving performance during the physical completion of given tasks.Because training in MI is relatively easy and effective in improving motor performance, it has recently been used to improve motor deficits in stroke and Parkinson's disease. Due to the severe motor impairments in pwMS and the negative effects of these impairments on QoL, it has recently been recommended for therapeutic use in MS. A study found that patients with MS had significant differences in the mean accuracy and temporal organization of MI ability compared to age-matched healthy controls.

MI skills are associated with motor planning and regulation.Studies have shown that cognitive performance measured by processing speed and executive function is significantly related to patients' motor function. In one study, the MI ability of pwMS differed significantly in the mean accuracy and temporal organization of MI compared to the MI ability of age-matched healthy controls.

Health-related QoL is an individual's assessment of how a health problem and its treatment affect the ability to perform daily life activities and roles. Studies have shown that pwMS report lower QoL than healthy controls or those with other chronic diseases such as rheumatoid arthritis and inflammatory bowel disease.

There is no study evaluating upper extremity MI skills in pwMS and examining its effects on upper extremity functional skills and QoL. In this direction, the aim of this study is to investigate the relationship between upper extremity MI ability and upper extremity functional skills and QoL in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older
* Mini Mental Test score of 24 or higher
* No neuro-musculoskeletal disease

Exclusion Criteria:

* Being pregnant
* Having a neuromusculoskeletal disease other than Multiple Sclerosis
* Having any contractures in the upper extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Have a confirmed MS diagnosis according to the revised McDonald criteria
  * Be 18 years of age or older
  * Have a Mini Mental Test score of 24 or higher
  * Have not changed medication in the last 6 months
  * Have not had an attack in the last 3 months
  Exclusion Criteria:
  * Being pregnant
  * Having a neuromusculoskeletal disease other than Multiple Sclerosis
  * Having any contractures in the upper extremity
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
The Kinesthetic and Visual Imagery Questionnaire (KVIQ) | 1st day of the interview
  It was created by Malouin and his colleagues in 2007 based on the KVIQ to assess the kinesthetic and visual imagery abilities of healthy and physically disabled individuals. The movements in the items in the questionnaire are first physically performed by the individual and then the same movement is imagined. The clarity of visual imagery and the intensity of kinesthetic imagery are scored on a 5-point scale. Since the Kinesthetic and Visual Imagery Questionnaire includes simple movements performed while sitting, it was developed for individuals who cannot stand for various reasons, cannot perform complex movements, and need guidance during imagery. A higher score indicates better kinesthetic perception. Minimum score is 20 and maxmum score is 100.
Mental Stopwatch | 1st day of the interview
  Mental chronometry is based on comparing the time taken to perform a movement with the time taken to image the same movement. The score obtained from mental chronometry can be affected by various factors such as the duration of the activity, complexity, type of motor imagery (kinesthetic or visual) and the instructions given. Mental chronometry is related to the individual's ability to maintain and control the imaged image. Mental chronometry is based on the comparison between the physical execution time of a task and the imagined one, with a close temporal relationship indicating correct MI. In our study, DDPT will be used as the mental chronometry evaluation method due to its practicality and accessibility.
Nine Hole Peg Test (NHPT) | 1st day of the interview
  It was first introduced by Kellor et al. in 1971. During the test, the patient sits at a table with a 9-hole board in front of him, inserts and removes wooden or plastic rods into 9 empty holes. The insertion and removal times are recorded. The test is performed 3 times in succession for the dominant hand and the non-dominant hand. The test score is the average of these three trials. In our study, the NHPT will be applied as a mental stopwatch test. In the application part, after a practice trial, three physical applications and three motor imagery trials will be performed for each hand, respectively. During the imagery trials, participants will be instructed to use visual images from a first-person perspective and will be asked to imagine performing the same task physically. The average time of these three physical applications and imagery trials for both hands will be calculated and recorded.
Jebson-Taylor Hand Function Test (JTHFT) | 1st day of the interview1
  It was developed in 1969 to evaluate the effectiveness of treatment and disability in patients with hand injuries. The JTHFT consists of tasks aimed at evaluating a wide range of one-handed hand functions required for daily living activities. The 7 test items required to be performed must be repeated for both hands. The functions of both hands are evaluated with the following operations; writing, turning over 8x13 cm paper cards, picking up small objects, simulating eating, stacking backgammon-checker checkers, picking up large objects, picking up large and heavy objects. The completion time of each task is recorded separately. The tasks are performed using both hands, first the non-dominant hand. The total application time of the test is around 45 minutes.
Manual Ability Measure-36 (MAM-36) | 1st day of the interview
  MAM-36 has been used to assess subjective upper extremity function in people with a variety of neurological and non-neurological diseases. Additionally, the MAM-36 is one of the most commonly used patient-reported outcome measures in patients with multiple sclerosis (pwMS). The MAM-36 contains 36 items asking about the perceived ease or difficulty of performing common tasks; rated on a 4-point Likert-type scale from 0 (almost not performed) to 4 (easy).Higher MAM-36 scores indicate higher functional ability.
multiple sclerosis impact scale-29 | 1st day of the interview
  It is a scale that evaluates the quality of life in MS patients, developed by Hobart et al. in 2001. It contains 20 statements covering physical parameters related to MS disease and a 9-item statement covering psychological problems. The physical section includes items from 1 to 20. The psychological section is ranked from 21 to 29. Participants are asked to answer each item regarding the impact of the condition on their daily lives in the last two weeks. Patients select the response that most strongly represents their condition and respond to each item on a 5-point Likert scale. The patient's scores on the two subscales can be added and converted to a measurement between 0 and 100. Higher scores indicate higher disease impact.

SECONDARY OUTCOMES:
Expanded disability status scale (EDSS) | 1st day of the interview
  It is used to determine the degree of neurological disability in individuals with MS and determines their functional capacity. It evaluates the functions of eight functional systems of the Central Nervous System (pyramidal, cerebral, brainstem, vision, bladder and bowel, sensory and cerebral). Each of these systems is scored according to the severity of the impairment in their functions. After the limitations in daily life are added to these functional system scores, an EDSS score ranging from 0 to 10 is obtained. The EDSS scores to be used in our study will be obtained from the clinical reports of the physician who follows the patient.
Mini-Mental State Examination (MMSE) | 1st day of the interview
  The test was produced as a short-term cognitive assessment tool to quantitatively evaluate cognitive performance within standard neuropsychiatric examination methods. Although the test has limited specificity in terms of distinguishing clinical syndromes, it is a short, practical and standardized method that can be used to determine the global cognitive level. It consists of eleven items grouped under five main headings: orientation, recording memory, attention and calculation, recall and language, and is evaluated out of a total score of 30. A score of 24 and above is determined as normal. A Turkish validity and reliability study has been conducted (27). Since MMSE is an inclusion criterion, it will be applied to participants while recruiting them to the study.
Fatigue Severity Scale (FSS) | 1st day of the interview
  It is a scale developed to measure the severity of fatigue and is widely used in individuals with MS, with high reliability and validity. The scale questions the severity of fatigue in the last month. The scale consists of 9 questions and each question is graded out of 7 points. A score of 28 and above is the fatigue limit, and a high score indicates more fatigue. The scale has been validated and reliable in Turkish in individuals with MS. The purpose of using FSS in our study is that fatigue is an important symptom in MS and is supported by studies in the literature that it affects motor imagery ability.
Beck Depression Inventory (BDI) | 1st day of the interview
  The Beck Depression Inventory, or inventory as it is also known, was developed by Beck and his colleagues in 1961 and is a scale that evaluates the characteristic features and symptoms of depression. Since its development, different versions have been released with various updates. The scale is a self-report scale. It does not require a clinician to administer it. It consists of 21 items and takes approximately 10 minutes to complete. Each item is a multiple choice between 0 and 3. The person marks the option that best describes them. Then, the score given to each item is added up. The lowest score that can be obtained from the scale is 0, and the highest score is 63. According to the total score obtained; it is concluded that it is none-mild, mild-moderate, moderate-severe or severe. Emotional symptoms such as depression are common in MS patients and it has been stated in the literature that they affect motor imagery ability.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozkeskin, Pt, PhD, Study Director — Ege University
Locations (1):
- Hatice Adiguzel, Kahramanmaraş, Onikisubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No